CLINICAL TRIAL: NCT05729724
Title: Effect of Pharmacological Interventions Aimed to Increase Arterial Blood Pressure on Systolic Blood Pressure Drops Evidenced by 24-hour Ambulatory Blood Pressure Monitoring in Patients With Reflex Syncope
Brief Title: Effect of Pharmacological Interventions on Systolic Blood Pressure Drops (SynABPM 2 Proof-of-concept)
Acronym: SynABPM
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C216
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Syncope; Syncope, Vasovagal; Ambulatory Blood Pressure Monitoring; Antihypertensive Drugs; Orthostatic Hypotension
Keywords: Syncope; Tilt testing; Carotid sinus massage; 24-hour ABPM
MeSH Terms: conditions — Syncope; Syncope, Vasovagal; Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Change treatment: Deprescribing (patients on hypotensive medications): withdrawal or reduction of one or more medications among cardiovascular and psychoactive drugs with known hypotensive effects (Table) Prescription of vasoactive medications (patients with constitutional hypotension): prescription of Fludrocortisone or other drugs that actively increase blood pressure.

SUMMARY:
SynABPM 2 proof-of-efficacy is a retrospective, multicentre, observational study performed in patients affected by hypotensive reflex syncope who had performed two ABPMs, one before and another after any therapeutical intervention aimed to increase arterial blood pressure

DETAILED DESCRIPTION:
24-hour ambulatory blood pressure monitoring (ABPM) is able to detect systolic blood pressure (SBP) drops that allow to discriminate patients with reflex syncope from controls. One episode of daytime SBP <90 mmHg or one episode of daytime SBP <100 mmHg, if mean 24-hour SBP is <125 mmHg, is the best cut-off for the identification of reflex syncope patients with hypotensive susceptibility.

The hypothesis of the present proof-of-concept study is that a therapeutic strategy aimed to increase arterial blood pressure can prevent SBP drops and (hopefully) reduce syncope recurrences.

If the study hypothesis will be confirmed, the magnitude of increase of SBP needed to abolish SBP drops will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were those who fulfilled all the following criteria:

* had received a diagnosis of reflex syncope
* had undergone an ABPM as part of the routine work-up of syncope in use in these hospitals that had shown one or more daytime SBP drop <90 mmHg or one or more daytime drops <100 mmHg in patients with average 24-hour SBP ≥125 mmHg
* had received instructions in order to abolish/reduce their antihypertensive therapy with the aim to prevent syncopal recurrences or had received active drug therapy, i.e., fludrocortisone, in order to increase their arterial blood pressure.
* had performed a second ABPM within 6 months from ABPM 1 in order to verify the effect of the prescribed change in therapy

Exclusion Criteria:

* Age <18 years
* Symptomatic orthostatic hypotension (defined as a symptomatic fall in SBP ≥20 mm Hg or a SBP decrease to <90 mmHg, as per the ESC guidelines;
* competing causes of syncope (i.e., syncope due to arrhythmias and structural cardiac diseases and non-syncopal causes of transient loss of consciousness as defined by ESC guidelines on syncope
* Severe structural heart disease, previous stroke or transient ischaemic attack

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by hypotensive reflex syncope who had performed two ABPMs, one before and another after any therapeutical intervention aimed to increase arterial blood pressure
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation | two months
  Correlation between changes in 24-hour average SBP and burden of SBP drops

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the study
Access Criteria: mbrignole@outlook.it

REFERENCES:
- [Background] Rivasi G, Groppelli A, Brignole M, Soranna D, Zambon A, Bilo G, Pengo M, Sharad B, Hamrefors V, Rafanelli M, Testa GD, Rice C, Kenny RA, Sutton R, Ungar A, Fedorowski A, Parati G. Association between hypotension during 24 h ambulatory blood pressure monitoring and reflex syncope: the SynABPM 1 study. Eur Heart J. 2022 Oct 11;43(38):3765-3776. doi: 10.1093/eurheartj/ehac347. PMID 35766175
- [Derived] Groppelli A, Rivasi G, Fedorowski A, de Lange FJ, Russo V, Maggi R, Capacci M, Nawaz S, Comune A, Bianchi L, Zambon A, Soranna D, Ungar A, Parati G, Brignole M. Interventions aimed to increase average 24-h systolic blood pressure reduce blood pressure drops in patients with reflex syncope and orthostatic intolerance. Europace. 2024 Feb 1;26(2):euae026. doi: 10.1093/europace/euae026. PMID 38262617